CLINICAL TRIAL: NCT02522364
Title: Subclinical Postoperative Atrial Fibrillation
Acronym: POAF-ILR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Michael Glikson, Director of Davidai Arrhythmia Center, Leviev Heart Center, Sheba Medical Center, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SHEBA-05-2282-MG-CTIL
Record Dates: First submitted 2015-07-28; First posted 2015-08-13 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Atrial Fibrillation
Keywords: Postoperative atrial fibrillation; Dysfunction Following Cardiac Surgery
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BioMonitor (Active Comparator): Participants randomized for this arm will be implanted with a BioMonitor device an implantable loop recorder inserted under the skin in the region of the thorax. It continuously records heart rhythm for a period of up to 7 years. The device will be interrogated at 1 month intervals. All arrhythmic events and conductive disturbances will be noted. In addition will be followed as specified in the standard arm
  Interventions: Device: BioMonitor device
- Standard (Active Comparator): Participants randomized for this arm will be followed by biannual office visits initialing clinical evaluation, review of clinical events, review and update of medical therapy. Participants will undergo ECG holter examination at 3 and 6 months after discharge
  Interventions: Other: Standard

INTERVENTIONS:
Device: BioMonitor device — Implantation of a BioMonitor device and continuously monitoring heart rhythm for study duration
  Arms: BioMonitor
Other: Standard — Clinical and intermittent electrocardiographic follow-up of patients
  Arms: Standard

SUMMARY:
Postoperative atrial fibrillation and atrial flutter (POAF) is the most common complication after cardiac surgery requiring intervention or prolonged hospital stay.

POAF is associated with higher mortality and higher risk of thromboembolic events.

However, It is yet unknown whether a now event of postoperative atrial fibrillation is an indication of a chronic arrhythmic disease - a tendency towards developing recurrent atrial fibrillation or merely a response to the stress of surgery with not recurrence. This distinction is critical to determine the appropriate therapy. Since recurred events of atrial fibrillation (Paroxysmal atrial fibrillation) are associated with long term risk for stroke and thromboembolic evens patients with PAF are treated with long term anticoagulation. Missing the long term recurrence of arrhythmia may result in under-treatment and pose a significant risk of stroke.

Bio-Monitor is a subcutaneous implanted device that automatically detects arrhythmias and stores electrocardiogram (ECG) recordings. It will enable the detection of atrial fibrillation over a period of years and allow correct diagnosis and appropriate treatment.

The purpose of the study is to study the long term behavior of POAF, determine the likelihood of developing paroxysmal atrial fibrillation in patients with POAF and to define the risk factors for this eventuality

DETAILED DESCRIPTION:
Clinical background:

Postoperative atrial fibrillation and atrial flutter (POAF) is the most common complication after cardiac surgery requiring intervention or prolonged hospital stay . Affecting 10-65% of patients , this arrhythmia is associated with increased mortality, considerable morbidity including systemic therombo-embolism and hemodynamic deterioration. Often it will prolong the hospital stay and increase health costs. Notably, the incidences of POAF is increasing resulting from an increase in the average age and arrhythmic risk factors in patients undergoing cardiac surgery.

Although a lot of POAFs occur in patients with a history of PAF, there is an important portion of POAF in patients who have never experienced AF before. In some of these patients POAF may be the first manifestation of a tendency to fibrillate (that may have been silent prior to surgery) whereas in others it may be an acute response to the peri-operative stress that may never recur after the acute phase. A recent study has shown that patients with a first detected AF episode precipitated by a secondary event (the most common of which was cardiothoracic surgery) are very likely to have recurrent events. In fact the risk of recurrence was similar to that of patients with an AF event with an obvious precipitating factor Current guidelines mainly address the acute management of arrhythmia. Most conclude that anti-thrombotic therapy is indicated in POAF (IIA) usually if the arrhythmia persists for at least 48 hours. However this recommendation is based on very limited evidence as there is no substantial data describing the long term natural history of this complication. POAF was described as self-terminating but frequently recurrent with a complete resolution within 6-12 weeks . However, this observation was based on electrocardiogram follow-up with no continuous long term monitoring (ECG holter or loop recorder) and are therefore of limited validity. Emerging data suggests that AF recurrence rates may be significate ranging up to 24% over 6 years . Still, it is currently unknown how many of the patients presenting with an acute episode of POAF will develop recurrent events and when, as a result, there are no clear recommendations regarding the duration of anticoagulantion treatment. The current practice in cases of POAF of significant duration is to administer anti-coagulation therapy combined with antiarrhythmic (most often with amiodarone) for 6-12 weeks. The only guideline based recommendation that is based on poor evidence is to administer OAC to AF patients following CABG for at least 3 months . Holter ECG is routinely performed prior to the end of this period and if normal and clinical evaluation is normal the treatment is discontinued, usually with no additional evaluation.

Technical overview:

This study will be executed using the following devices and services:

* BioMonitor is a subcutaneous implanted device that automatically detects arrhythmias and stores electrocardiogram (ECG) recordings. It is implanted in a small subcutaneous pocket, similar to a pacemaker but without the need for inserting electrodes. It provides high quality ECG recording and has longevity of 6.4 years. In addition it has wireless capabilities and may transmit data to an external modem (CardioMessenger) and though it to an internet based network - the Home-Monitoring.
* HomeMonitoring is an Internet-based, automatic, remote, monitoring system that uses the cellular phone network to enable transmissions of recorded data and alerts from the HM Service Center to a predefined email address, fax or a cellular phone.

Study propose The investigators hypothesize that the intermediate and long term burden of newly diagnosed POAF is significantly greater than currently described. We further hypothesize that it may be a marker for affected atria representing a greater risk for chronic arrhythmia. Therefore, we believe that a substantial group of patients presenting with POAF will have atrial fibrillation recurrences (paroxysmal, persistent or permanent) requiring long term anticoagulation We also believe that with the help of ILR we will be able define a subgroup of POAF patients in whom POAF is related to the acute phase and are not prone to recurrence nor do they need long term anticoagulation In this pilot study we propose to use an ILR to diagnose both symptomathic and asymptomatic events of atrial fibrillation in subjects after cardiac surgery. We intend to define the natural history of post-operative atrial fibrillation and to identify the predictors for recurrent events.

Study aims:

1. To evaluate the incidence of recurrent AF events, during long term follow-up in patients presenting with newly diagnosed POAF discharged in sinus rhythm.
2. To identify predictors for the development of recurrent AF events
3. To verify the use of implantable loop recorders (ILRs) as tools in detection of AF and anticoagulant management in POAF
4. To evaluate rates of mortality and major adverse events (CVA, systemic thromboembolism, rapid AF requiring hospitalization) among patients presenting with POAF discharged in sinus rhythm.
5. To identify predictors for mortality and major adverse events.

Methods - general Study design - pilot

• A multicenter, prospective randomized, open label interventional study

* Participants will be randomized in a ratio of 2:1 to implantation of loop recorder or usual follow up
* Participants will be followed for a median of 2 years.
* Country of primary site - Israel Study population
* Participants will be recruited from patients admitted to a cardiac surgery ward in participating medical centers
* Participants will be recruited during index hospitalization or within a week after discharge Recruitment & randomization

  1. Requirement will begin on the 1st of August 2015
  2. Potential participants will receive a comprehensive explanation.
  3. All participants will sign an informed consent form
  4. A baseline CRF will be filled (see appendix A1)
  5. Baseline evaluation a. Medical interview and review of electronic patient file b. physical examination c. ECG- 12 lead test at recruitment d. Laboratory test - CBC, Chemistry including electrolytes, kidney and liver function
  6. Randomization

     1. Will be performed at the time of requirement
     2. Will be carried out by using standard software Device & device implantation

  1. Device

  a. The1st generation Biomonitor device will be used in this study b. Arrhythmia detection based on R-R interval analysis c. The device will identify and record the following rhythms automatically: i. Asystole - R-R interval >5 sec ii. Bradycardia / sudden rate drop - rate<40 BPM for >20 seconds (options: 5, 10, 15, 25 or 30 sec) OK iii. Atrial Fibrillation -
  1. AF Sensitivity - Medium
  2. R-R interval variability - 12.5%
  3. Onset/Resolution window - 8/16
  4. AF onset intervals - 5
  5. AF resolution intervals - 1
  6. Confirmation time - 5 minutes
  7. AF termination criteria - 5/8intervals iv. High ventricular rates - rate>180 BPM for >16 beats d. The device will allow for patient activated recording. e. Automatically detected events will be recorded for 40 sec (30 sec pre and 10 sec of the events) and 7.5 minutes of patient activated events (7 min pre and 30 sec post activation).

     f. The duration of each arrhythmic event will be recorded. g. ECG tracings of each type of event will be stored

  2. Device implantation
  1. ILR will be inserted during index hospitalization
  2. Apixaban will we withheld according to EHRA NOAC document as related to renal function prior to device implantation and will be resumed 48 hours after it's completion
  3. For patients on VKA The implantation will be postponed if INR at the day of the procedure exceeds 3
  4. The device will be implanted in a tight pre-pectoral pocket.
  5. Device location will be defined by implanting physician based on signal quality.
  6. Prophylactic antibiotic treatment will be given both before and after implantation. The antibiotic agents will be selected according the protocol designed for pacemaker implantation in the various centers.
  7. An implantation CRF will be filled upon completion of procedure (appendix A1)

     Pre-discharge recommendations

     1. Implantation site will be examined by a trained physician 2. All participants will undergo a standard echocardiography .Test results will be evaluated by a core lab 3. Results of the examination will be noted on CRF

     Discharge recommendations 1. All patients will be discharged on OAC for three months (according to ESC revascularization guidelines )

  a. Patients with valvular (significant and uncorrected mitral stenosis) disease will be treated with warfarin b. Patients with no valvular disease will be treated with apixaban 2. These will be stopped after 90 days without AF according to the assigned follow up method as long as no more than 120 days elapsed since hospital discharge 3. If AF of more than 5 minutes recurs anticoagulation will be continued active or resumed if already discontinued.

  4. A recommendation for an anti-arrhythmic agent, for duration of a maximum of 6 weeks will be left to the discretion of the attending physician.

  5. Continuation of anti-arrhythmic therapy will be done only in cases of clinical and symptomatic AF Follow-up
  1. Clinical follow-up - Biannual office visits

     a. Participants will be asked to report any relevant symptoms or clinical events including hospitalizations, CVA/TIA, events of syncope, pre-syncope, overt atrial fibrillation, palpitations or chest discomfort b. Active medical therapy will be updated c. All data will be recorded in the clinical follow-up CRF (appendix B1)
  2. ECG monitoring

     a. BioMonitor i. The ILR will be interrogated at 1 month intervals ii. The quality and integrity of ECG tracings will be evaluated at each visit and the device's programing will be updated by the core lab to overcome under-sensing, T-wave over-sensing or other misdiagnosis.

     b. Home Monitoring system - optional preferable i. Study participants will be supplied with a CardioMessenger unit ii. The BioMonitor will transmit relevant event data on a daily basis iii. Continuouss monitoring will be done through the Home Monitoring system iv. Event log will be reviewed by the attending physician on every two days c. EGC holter i. Participants will undergo ECG holter examination at 3 and 6 months after discharge d. All data will be recorded in the clinical ECG event log CRF (appendix B2)
  3. Laboratory follow-up - Routine CBC once every 6 months

ELIGIBILITY:
Inclusion Criteria:

* Newly documented POAF of more than 5 minute duration
* cardiac surgery during index hospitalization, including (CABG, valvular replacement or repair, a combination) without Maze procedure
* CHA2DS2-VASc≥2
* Sinus rhythm at the time of BioMonitor implantation or definite intention to cardiovert prior to discharge
* Signed Informed Consent

Exclusion Criteria:

* History of atrial fibrillation/flutter prior to cardiac surgery
* Contraindication for anticoagulation therapy
* Dual chamber pacemaker or ICD implanted or planned
* Active systemic infection
* Another (non-AF) indication for long term anticoagulation
* Maze procedure
* Inability to attend scheduled, periodic office visits for follow-up
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation event | 2 years
  Documented Atrial fibrillation of more the 5 minutes duration
MACCE | 2 years
  A composite of all -cause mortality, CT/MRI proven stroke, CT proven systemic embolism
Implantation of permanent pacemaker | 2 years
Implantation of ICD | 2 years
  Implantation of ICD following documented ventricular arrhythmia
Pocket hematoma | 30 days
  The development of a hematoma in the BioMonitor insertion site
Pocket site infection | 2 years
  The development of a Pocket site infection in the BioMonitor insertion site
Device extraction | 2 years
Major bleeding | 2 years
  A composite of the following events:
  i. Bleeding resulting in a decrease in hemoglobin of ≥2 g/dL or over a 24-hour period ii. Bleeding leading to a transfusion of 2 or more units of packed red blood cells iii. Bleeding that occurs in a critical site (intracranial, intraspinal, intraocular, pericardial, intra-articular, intramuscular with compartment syndrome or retroperitoneal) iv. Bleeding that leads to death.

SECONDARY OUTCOMES:
All -cause mortality | 2 years
CT/MRI proven stroke | 2 years
Rapid AF requiring hospitalization | 2 years
Initiation of long term anti-coagulation therapy | 2 years
Initiation of long term anti-arrhythmic therapy | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Glikson, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

REFERENCES:
- [Result] Aranki SF, Shaw DP, Adams DH, Rizzo RJ, Couper GS, VanderVliet M, Collins JJ Jr, Cohn LH, Burstin HR. Predictors of atrial fibrillation after coronary artery surgery. Current trends and impact on hospital resources. Circulation. 1996 Aug 1;94(3):390-7. doi: 10.1161/01.cir.94.3.390. PMID 8759081
- [Result] Mitchell LB; CCS Atrial Fibrillation Guidelines Committee. Canadian Cardiovascular Society atrial fibrillation guidelines 2010: prevention and treatment of atrial fibrillation following cardiac surgery. Can J Cardiol. 2011 Jan-Feb;27(1):91-7. doi: 10.1016/j.cjca.2010.11.005. PMID 21329866
- [Result] Maisel WH, Rawn JD, Stevenson WG. Atrial fibrillation after cardiac surgery. Ann Intern Med. 2001 Dec 18;135(12):1061-73. doi: 10.7326/0003-4819-135-12-200112180-00010. PMID 11747385
- [Result] Creswell LL, Schuessler RB, Rosenbloom M, Cox JL. Hazards of postoperative atrial arrhythmias. Ann Thorac Surg. 1993 Sep;56(3):539-49. doi: 10.1016/0003-4975(93)90894-n. PMID 8379728
- [Result] European Heart Rhythm Association; European Association for Cardio-Thoracic Surgery; Camm AJ, Kirchhof P, Lip GY, Schotten U, Savelieva I, Ernst S, Van Gelder IC, Al-Attar N, Hindricks G, Prendergast B, Heidbuchel H, Alfieri O, Angelini A, Atar D, Colonna P, De Caterina R, De Sutter J, Goette A, Gorenek B, Heldal M, Hohloser SH, Kolh P, Le Heuzey JY, Ponikowski P, Rutten FH. Guidelines for the management of atrial fibrillation: the Task Force for the Management of Atrial Fibrillation of the European Society of Cardiology (ESC). Eur Heart J. 2010 Oct;31(19):2369-429. doi: 10.1093/eurheartj/ehq278. Epub 2010 Aug 29. No abstract available. PMID 20802247
- [Result] January CT, Wann LS, Alpert JS, Calkins H, Cigarroa JE, Cleveland JC Jr, Conti JB, Ellinor PT, Ezekowitz MD, Field ME, Murray KT, Sacco RL, Stevenson WG, Tchou PJ, Tracy CM, Yancy CW; ACC/AHA Task Force Members. 2014 AHA/ACC/HRS guideline for the management of patients with atrial fibrillation: executive summary: a report of the American College of Cardiology/American Heart Association Task Force on practice guidelines and the Heart Rhythm Society. Circulation. 2014 Dec 2;130(23):2071-104. doi: 10.1161/CIR.0000000000000040. Epub 2014 Mar 28. No abstract available. PMID 24682348
- [Result] Kowey PR, Stebbins D, Igidbashian L, Goldman SM, Sutter FP, Rials SJ, Marinchak RA. Clinical outcome of patients who develop PAF after CABG surgery. Pacing Clin Electrophysiol. 2001 Feb;24(2):191-3. doi: 10.1046/j.1460-9592.2001.00191.x. PMID 11270698
- [Result] Lee JK, Klein GJ, Krahn AD, Yee R, Zarnke K, Simpson C, Skanes A, Spindler B. Rate-control versus conversion strategy in postoperative atrial fibrillation: a prospective, randomized pilot study. Am Heart J. 2000 Dec;140(6):871-7. doi: 10.1067/mhj.2000.111104. PMID 11099990
- [Result] Pillarisetti J, Patel A, Bommana S, Guda R, Falbe J, Zorn GT, Muehlebach G, Vacek J, Sue Min Lai, Lakkireddy D. Atrial fibrillation following open heart surgery: long-term incidence and prognosis. J Interv Card Electrophysiol. 2014 Jan;39(1):69-75. doi: 10.1007/s10840-013-9830-6. Epub 2013 Nov 29. PMID 24293173
- [Result] Ahlsson A, Fengsrud E, Bodin L, Englund A. Postoperative atrial fibrillation in patients undergoing aortocoronary bypass surgery carries an eightfold risk of future atrial fibrillation and a doubled cardiovascular mortality. Eur J Cardiothorac Surg. 2010 Jun;37(6):1353-9. doi: 10.1016/j.ejcts.2009.12.033. PMID 20138531
- [Result] Authors/Task Force members; Windecker S, Kolh P, Alfonso F, Collet JP, Cremer J, Falk V, Filippatos G, Hamm C, Head SJ, Juni P, Kappetein AP, Kastrati A, Knuuti J, Landmesser U, Laufer G, Neumann FJ, Richter DJ, Schauerte P, Sousa Uva M, Stefanini GG, Taggart DP, Torracca L, Valgimigli M, Wijns W, Witkowski A. 2014 ESC/EACTS Guidelines on myocardial revascularization: The Task Force on Myocardial Revascularization of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS)Developed with the special contribution of the European Association of Percutaneous Cardiovascular Interventions (EAPCI). Eur Heart J. 2014 Oct 1;35(37):2541-619. doi: 10.1093/eurheartj/ehu278. Epub 2014 Aug 29. No abstract available. PMID 25173339
- [Result] Lee SH, Kang DR, Uhm JS, Shim J, Sung JH, Kim JY, Pak HN, Lee MH, Joung B. New-onset atrial fibrillation predicts long-term newly developed atrial fibrillation after coronary artery bypass graft. Am Heart J. 2014 Apr;167(4):593-600.e1. doi: 10.1016/j.ahj.2013.12.010. Epub 2014 Jan 4. PMID 24655710
- [Result] Lubitz SA, Yin X, Rienstra M, Schnabel RB, Walkey AJ, Magnani JW, Rahman F, McManus DD, Tadros TM, Levy D, Vasan RS, Larson MG, Ellinor PT, Benjamin EJ. Long-term outcomes of secondary atrial fibrillation in the community: the Framingham Heart Study. Circulation. 2015 May 12;131(19):1648-55. doi: 10.1161/CIRCULATIONAHA.114.014058. Epub 2015 Mar 13. PMID 25769640